CLINICAL TRIAL: NCT01213303
Title: Relation Between Fatty Acids and Oxidative Stress Markers With Cardiovascular Risk Factors in a Healthy Population
Brief Title: Cardiovascular Risk Factors, Lipid Metabolism and Oxidative Stress
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Luigi Iuliano, M.D., University of Roma La Sapienza
Other Study IDs: Iuliano_AVIS
Record Dates: First submitted 2010-09-30; First posted 2010-10-01 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Cardiovascular Disease
Keywords: cardiovascular risk; metabolic syndrome; fatty acids; oxysterols; antioxidants; oxidative stress
MeSH Terms: conditions — Cardiovascular Diseases; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples Without DNA — Collection of plasma and serum samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Blood donors: Evaluation of cardiovascular risk factors, oxidative stress and fatty acid metabolism in a cohort of blood donors

SUMMARY:
Cardiovascular diseases belong to the major causes of mortality in western populations, and atherosclerosis is the lesion responsible for clinical events, such as acute myocardial infarction and stroke.

Atherosclerosis remains asymptomatic until a clinical event occurs, and in the pre-clinical stage it may be difficult to diagnose. As disease surrogate, a large number of risk factors for atherosclerosis are being recognized. Some of them are responsible for the epidemiologically very serious metabolic syndrome, which accounts for development of hyperlipidemia, obesity, diabetes or arterial hypertension.

Health providers in continental diet-based countries suggest to embracing Mediterranean diet in order to contribute in reducing cardiovascular mortality. However, countries in the Mediterranean area are experiencing a shift in dietary habit towards continental diet with potential harmful change in mortality rates. Oxidative stress, including free radical-driven reactions and antioxidant status are considered important mediators to be considered in the diet-mediated effect on health. Important metabolic functions are also mediated by certain fatty acids. A comprehensive study of oxidative stress, including free radical-driven products and protective antioxidants, and fatty acids metabolism has never been reported in healthy subjects. In particular, high sensitive mass-spectrometry methods to study oxidative stress and fatty acids metabolism are rarely applied to epidemiological studies.

The aim of the present grant project is therefore to assess in a large cross-sectional study the prevalence of oxidative stress markers, and fatty acids and to find any causal relation between these variables and metabolic syndrome. This population sample will be followed prospectively not only for time of the present grant project, but we would like to study metabolic variables with relation to the development of oxidative stress-mediated diseases, in particular those of cardiovascular system, on a longitudinal basis (prospective epidemiological study for at least 10 years). At same time we should be able to define the importance of individual markers of oxidative stress and fatty acids for early detection of these diseases.

DETAILED DESCRIPTION:
Background Cardiovascular diseases belong to the major causes of mortality in western populations. Atherosclerosis of arterial system may result in ischemic heart disease (IHD) and peripheral artery disease with possible fatal consequences such as acute myocardial infarction and stroke.

Atherosclerosis is a chronic and slowly growing pathological lesion that remains asymptomatic until a clinical event occurs. In the pre-clinical stage atherosclerosis may be difficult to diagnose. As disease surrogate, a large number of risk factors for atherosclerosis are being recognized. Some of them are responsible for the epidemiologically very serious metabolic syndrome, which accounts for development of hyperlipidemia (from preventive point of view only 25% of population has normal blood lipid levels), obesity, diabetes or arterial hypertension. In all of these conditions, oxidative stress represents a substantial pathogenic factor through deleterious chemical reactions that damage biomolecules, including formation of atherogenic- oxidatively-modified LDL particles (1) or direct destruction of cells and tissues by free radicals (2-4). Lifestyle, in particular dietary schemes, belongs to important factors contributing to the formation and development of atherosclerosis. The usefulness of dietary components in contributing to low cardiovascular mortality in populations of the mediterranean basin is well recognized. After pioneering studies by Ancel Keys (5), Mediterranean diet has become popular worldwide as health diet. Several components of this diet have been advocated in contributing to counteract atherosclerosis, including a panel of antioxidants and unsaturated fatty acids. Health providers in continental diet-based countries suggest to embracing Mediterranean diet in order to contribute in reducing cardiovascular mortality. However, countries in the Mediterranean area are experiencing a shift in dietary habit towards continental diet with potential harmful change in mortality rates. Recently, Trichopoulou et al. (6) reported on adherence to mediterranean diet and survival in a Greek population. These authors found that adherence to this diet is associated with a significant reduction in mortality.

Italy is being challenged in lifestyle and dietary habit issues because such a drift has already caused an increase in obesity prevalence in children. Paradoxically, this is much higher in the south of Italy that is expected to be more strictly associated with mediterranean style.

It is not known, however, which components of the Mediterranean diet act protectively in the organism. It is suggested that certain components of the diet may importantly affect oxidative stress (7) and thereby also occurrence of cardiovascular (8) and tumor diseases (9). There are also very interesting data on the relation between regional dietary habits and diet composition, and the occurrence of cardiovascular diseases. From this point of view Mediterranean region seems to be exemplary. Low incidence of cardiovascular diseases was demonstrated here already in 50´s in spite of relatively high fat intake, whose major source was, however, olive oil rich in monounsaturated fatty acids and antioxidants such as polyphenolic compounds 12(10). Mediterranean diet was proved also in controlled studies to have marked protective effects on development of cardiovascular diseases (11, 12), but also total mortality (6) probably by action of antioxidant substances increasing total antioxidant capacity (13). The role of dietary factors on total antioxidant status was described in numerous studies, which showed marked increase of antioxidant potential after administration of vitamin A (14), vitamin C (15), tomatoes or tomato products containing high amounts of antioxidative terpen lycopene or lycopene together with olive oil (16).

On the other hand, it is emerging that previously unrecognized products of lipid metabolism may have profound effects on metabolic syndrome and potentially on the induction of diabetes. Palmitoleate has been recognized as an adipose-tissue derived lipid hormone that strongly stimulates muscle insulin action and suppresses hepatosteatosis (17). If palmitoleate acts as a lipid hormone in human is not known. In human, other fatty acids have been demonstrated to be altered in clinical conditions opposite to obesity. In fact, in cystic fibrosis patients, who are usually malnourished, we detected an increase in saturated and monounsaturated fatty acids (18) and a decrease in n-6 polyunsaturated fatty acids. C24:0 was positively correlated with BMI, plasma cholesterol and vitamin E, and significantly negatively correlated with oxysterols.Taken together, these data possibly identifies C24:0 as an indicator of adequate nutriture, coupled with the observation that C24:0 levels were reduced in patients with pancreatic insufficiency.

A comprehensive study of oxidative stress, including free radical-driven products and protective antioxidants, and fatty acids metabolism has never been reported in healthy subjects. In particular, high sensitive mass-spectrometry methods to study oxidative stress and fatty acids metabolism are rarely applied to epidemiological studies.

The aim of the present grant project is therefore to assess in a large cross-sectional study the prevalence of oxidative stress markers, and fatty acids and to find any causal relation between these variables and metabolic syndrome. This population sample will be followed prospectively to study metabolic variables with relation to the development of oxidative stress-mediated diseases, in particular those of cardiovascular system, on a longitudinal basis (prospective epidemiological study for at least 10 years). At same time we should be able to define the importance of individual markers of oxidative stress and fatty acids for early detection of these diseases.

During the time of proposed project, we want to examine, 500 healthy subjects divided in decade groups in the range between 20-60 years and in a group over 60 years. To do this we have identified a healthy cohort among blood donors. Blood donors are requested to be in healthy conditions but they are not devoid of cardiovascular risk factors, including metabolic syndrome.

Subjects will be informed in detail with the study proposal according to ethic principles and prior enrollment will sign informed consent.

In all examined subjects detailed medical history will be taken with special interest for diseases of cardiovascular system and risk factors for atherosclerosis. A complete physical exam including basic anthropometric examinations (BMI calculation and determination of waist circumference) and EKG will be performed in all subjects. Blood and urine collection will be performed to determine specific analytes:

1. Routine determinations - basic biochemistry (total cholesterol, HDL and LDL cholesterol, triglycerides, urea, creatinine, uric acid, glucose, AST, ALT, GMT, ALP, bilirubin),
2. Antioxidant vitamins in plasma - vitamins E, including α- and γ-tocopherol.
3. Markers of cholesterol oxidation (7β-hydroxycholesterol, 7keto-cholesterol) (determination by GC-MS)
4. Markers of arachidonate oxidation, F2 isoprostanes (determination by GC-MS)
5. Fatty acids profile (determination by GC-MS)

Since random population sample will be analyzed and measured variables will be determined on the continuous time scale, the above mentioned population sample (500 subjects) is sensitive enough to assess relations between metabolic syndrome and indicators of oxidative stress markers and lipid metabolism. Epidemiological approach (analysis of stratified data, linear and logistic regression, and statistical modelling of multipath relations) will be used to suppress the effect of confounding factors (e.g. age, smoking, sex) on data interpretation.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive enrollment of blood donors

Exclusion Criteria:

* Subjects with known chronic disease, including cardiovascular disease, liver disease, kidney disease, neurodegenerative disease and cancer; autoimmune disease, endocrine system disease,

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of healthy blood donors
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2009-05; Primary Completion 2015-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Fatty acids lipidomics and oxidative stress markers in healthy subjects | 21 months
  Assessment of plasma reference values of the complete fatty acid profile, oxysterols and alpha- and gamma-tocopherol in healthy italian subjects

SECONDARY OUTCOMES:
Prevalence of fatty acids levels, in a complete panel, and markers of oxidative stress in subjects with metabolic syndrome | 21 months
  The assessment of the complete fatty acids profile, oxysterols and vitamin E (alpha- and gamma-tocopherol) would reveal associations with components cardiovascular risk factors of the metabolic syndrome
Ten-year follow-up | ten years
  Prospective evaluation of cardiovascular events as function of baseline fatty acids and oxidative stress

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Iuliano, M.D., Ph.D., Study Director — University of Roma La Sapienza
Locations (2):
- Italy (2):
  - AVIS, Latina, Latina
  - Vascular Medicine Unit, Department of Medical Science and Biotechnology, Latina, Latina